CLINICAL TRIAL: NCT02140229
Title: REVECHO Study (REmission Véritable en ECHOgraphie) Is Ultrasound Remission a Real Remission? Does Ultrasound Permit to Achieve and Maintain the Remission in Rheumatoid Arthritis Patients More Efficiently Than Clinical Scores?
Brief Title: Is Ultrasound Remission a Real Remission? Does Ultrasound Permit to Achieve and Maintain the Remission in Rheumatoid Arthritis Patients More Efficiently Than Clinical Scores?
Acronym: REVECHO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P130401
Record Dates: First submitted 2014-05-07; First posted 2014-05-16 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Rheumatoid Arthritis; Remission
Keywords: Rheumatoid Arthritis; Remission,; DAS28,; ACR/EULAR,; RAPID, Randomized study,; Longitudinal follow-up
MeSH Terms: conditions — Arthritis, Rheumatoid; Fasting

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (Active Comparator): Usual care and follow-up every 3 months
  Interventions: Other: Usual care
- US-driven therapy (Experimental): Clinical evaluation according to DAS28 + US every 3 months
  Interventions: Device: US power doppler
- ACR/EULAR remission criteria-driven therapy (Active Comparator): Clinical evaluation according to DAS28 + ACR/EULAR remission criteria every 3 months
  Interventions: Other: ACR/EULAR criteria

INTERVENTIONS:
Device: US power doppler — Clinical evaluation according to DAS28 and US every 3 months. US examination is realized in B and Doppler power mode for each studied joint: Ankles, shoulders, elbows, wrists, MCP 1 to 5, PIP 1 to 5, knees and MTP 1 to 5.
  Arms: US-driven therapy
Other: Usual care — Clinical evaluation and follow-up according to the practice of the referring rheumatologist every 3 months
  Arms: Usual care
Other: ACR/EULAR criteria — Evaluation based on clinical evaluation according to DAS28 and ACR/EULAR remission criteria every 3 months.
  Arms: ACR/EULAR remission criteria-driven therapy

SUMMARY:
Remission is nowadays an achievable objective for Rheumatoid Arthritis (RA) patients thanks to a large choice of therapies, early treatment and tight control (30% relapse).

Ultrasound (US) driven-therapy, complemented with a clinico-biological follow-up, may improve the prognosis of RA in remission by increasing the duration of sustained remission and by preventing radiographic structural progression.

The tested hypothesis is: The US coverage of RA allows to increase the duration of sustained clinical remission.

DETAILED DESCRIPTION:
REVECHO is an international prospective multicentre simple blinded randomized study with a longitudinal follow-up of 18 months and a total study duration of 48 months. During the first visit, after having signed the consent form, Patients undergo at each visit, a clinical evaluation comprising an assessment of tender joint count (TJC), of swollen joint count (SJC), pain assessment, patient global assessment of the activity of disease, as well as a physician global assessment of the disease activity, an ultrasound examination of small and large joints by an independent physician blinded to the clinical data, and to the results of biological exams (blood sampling to assess CRP, complete blood count (CBS), and renal and hepatic functions). The clinical, biological and ultrasound assessments will be performed every 3 months.

Patients will be then randomly assigned to one of the 3 groups: 1) "Usual care group", 2) "Clinical (DAS28)-ultrasound follow-up group" (ultrasound-driven therapy) or 3) "DAS28-ACR/EULAR remission criteria group" (ACR/EULAR remission criteria-driven therapy), with a follow-up of 18 months.

Therapeutic decisions are taken by the Referring Rheumatologist. He/she will have DAS28 + US results in the group US follow-up or DAS28 + ACR/EULAR remission criteria results in the group ACR/EULAR follow-up. Therapeutic recommendations (therapeutic options, according to the randomization group, a threshold of activity will be decided by a scientific committee for increasing, stop or change therapy) will be given according to the group of randomization and based on the level of inflammation. The Referring Rheumatologist, will be free to follow or not the therapeutic advices.

In "Usual care" group, DAS28 and PDUS assessment will be performed at each time point, however, no suggestion neither DAS28 nor PDUS results will be given to the Referring Rheumatologist. The Referring Rheumatologist will be free to manage the patient as he/she thinks more appropriate.

Conventional radiography (hand and feet) will be performed at baseline and at M18 follow-up.

Centralized evaluation of radiographs will be performed by 2 independent readers, using SvH score. Radiographic progression will be defined by a change of SvH score between baseline and M18 >0.

PDUS examination will be performed every 3 months by an independent Physician in each centre, blinded to clinical, biological and radiographic data. Shoulders, elbows, wrists, MCP 1 to 5, PIP 1 to 5, knees, ankles (tibia-talar) and MTP 1 to 5 will be examined in B mode and in Power Doppler mode.

Each joint will be scored for synovitis according to the OMERACT definition and to the OMERACT scoring system (semi-quantitative score from 0 to 3 for grey scale, PD and for combined score).

Questionnaire (RAPID and HAQ) scores will be also evaluated every 3 months in each group.

ELIGIBILITY:
Inclusion Criteria:

1. RA patients (ACR 2010 criteria)
2. Disease duration ≤12 years
3. Patients of both genders above 18 years old
4. Remission according to DAS28 criteria (DAS28<2.6) since at least 3 months
5. Treated with DMARDS and/or biologics with stable posology since at least 3 months
6. Treated with corticosteroids ≤5 mg/day (oral, local intra-articular or perfusion) since at least 3 months
7. Affiliated to a regimen of health insurance (only for French sites)
8. Having signed a consent form
9. The patient is considered reliable, willing and capable of adhering to the protocol (for example, able to understand and complete diaries), visit schedule, and medication intake according to the judgment of the Investigator

Exclusion Criteria:

1. Pregnant women
2. Predictable difficulties of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time to loss of remission, as clinically defined by a DAS28 score ≥2.6 | Up to 18 months
  The DAS28 (Disease Activity Score for Rheumatoid Arthritis) score is calculated on the basis of swollen joint count (SJC) and tender joint count (TJC) out of 28 (shoulder, elbow, wrist, metacarpophalangeal (MCP) I-V, proximal interphalangeal (PIP) I-V, and knee) as follows:
  DAS28-CRP= 0.56 x √TJC + 0.28 x √SJC + 0.36 x Ln (CRP + 1) + 0.014 x GA + 0.96
  As a result, the DAS28 index gives a value between 0 and 10, with:
  * >5.1 indicating high disease activity
  * 3.2-5.1 indicating moderate disease activity
  * <3.2 indicating low disease activity
  * <2.6 complete remission

SECONDARY OUTCOMES:
Percentage of RA patients in clinical remission (DAS28 <2.6) at 18 months | 18 months
Percentage of RA patients without radiographic structural progression | 18 months
  Percentage of RA patients without radiographic structural progression (delta-Van der Heijde modified Sharp score ≤0) at 18 months.
Evolution of the RAPID score and HAQ | 18 months
  Evolution of the RAPID (Routine Assessment of Patient Index Data score) and HAQ (Health Assessment Questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Antonietta D'AGOSTINO, MD, PhD, Principal Investigator — Rheumatology Department, Ambroise Paré Hospital
Locations (1):
- Rheumatology Department, Ambroise Paré Hospital, Boulogne, Hauts DE Seine, France